CLINICAL TRIAL: NCT06895018
Title: Medium-term Effects of a Polyphenol-rich Beverage Based on Red Grape Pomace Extract on Non-alcoholic Fatty Liver Disease, Cardiometabolic Risk Profile and Gut Microbiota in Subjects with Type 2 Diabetes
Acronym: PoLiFat
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Giuseppina Costabile, Academic Researcher, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 325/20
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Polyphenols; NAFLD; Gut microbiota; Glucose metabolism; insulin metabolism; lipid metabolism; glucose variability; sublinical inflammation; grape pomace
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Grape Pomace Polyphenol Rich Drink (Experimental): Participants consume an experimental drink rich in polyphenols extracted from red grape pomace (RGP) containing 1.5 g/150 ml of Gallic Acid Equivalent (GAE) polyphenols and 28 g/150 ml of soluble sugars (14 g of glucose and 14 g of fructose) during the lunch and dinner for 6 weeks
  Interventions: Dietary Supplement: Supplementation with Polyphenol Rich Drink
- Placebo Drink (Placebo Comparator): Participants consume a control drink (Placebo), containing zero polyphenol and 28 g of total sugars (14 g of glucose and 14 g of fructose solubilized in 150 ml of drinking water), quantities equivalent to those contained in the experimental drink, during the lunch and dinner for 6 weeks
  Interventions: Dietary Supplement: Supplementation with Control Drink (Placebo)

INTERVENTIONS:
Dietary Supplement: Supplementation with Polyphenol Rich Drink — Participants were instructed to consume, over a 6-week period, within the context of a Mediterranean diet, a polyphenol-rich drink RGPD (150 mL) containing 1.5 g of polyphenols. After this treatment period, participants underwent a two-week washout period before switching to the alternative treatment with control drink (Placebo) devoid of polyphenols. To evaluate metabolic responses during both fasting and postprandial states, participants participants consumed a standardized test meal at the end of the 6 weeks. This standard meal was preceded by the consumption of the RGPD 60 minutes prior.
  Arms: Grape Pomace Polyphenol Rich Drink
Dietary Supplement: Supplementation with Control Drink (Placebo) — Participants were instructed to consume, over a 6-week period, within the context of a Mediterranean diet, a control drink (Placebo) (150 mL) containing 0 g of polyphenols. After this treatment period, participants underwent a two-week washout period before switching to the alternative treatment with a polyphenol-rich drink RGPD (150 mL) containing 1.5 g of polyphenols. To evaluate metabolic responses during both fasting and postprandial states, participants participants consumed a standardized test meal at the end of the 6 weeks. This standard meal was preceded by the consumption of the Control drink (Placebo) 60 minutes prior.
  Arms: Placebo Drink

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a liver disease characterized by an abnormal accumulation of fat not due to alcohol or drug consumption that can evolve into steatohepatitis (NASH), fibrosis and cirrhosis. Its prevalence is high, affecting approximately 20-30% of the general adult population and is also growing in pediatric age. Obesity, insulin resistance and type 2 diabetes (T2DM) are common and well-known risk factors for NAFLD, which is approximately 2-3 times more prevalent among obese and diabetic individuals. Despite the high and increasing prevalence of NAFLD in the population, its pathophysiology is not fully understood and there is currently no pharmacological treatment available.

Recent evidence suggests that dietary polyphenols may have specific beneficial effects on hepatic steatosis and associated sequelae by polyphenol metabolites and their phase II derivatives. Therefore, the aim of our study is to evaluate whether medium-term consumption of a beverage rich in polyphenols extracted from red grape pomace is able to exert beneficial effects on hepatic steatosis, cardiometabolic risk profile and microbiota composition of patients with type 2 diabetes.

DETAILED DESCRIPTION:
A randomized, crossover, placebo-controlled study will be conducted. Twenty patients with type 2 diabetes mellitus (T2DM) recruited from the Diabetes Unit of the University Hospital of Naples "Federico II" who meet the inclusion criteria will be studied. After a 2-week run-in period during which they will stabilize their habitual diet, participants will be randomly assigned to receive either 150 ml/day of a polyphenol-rich red grape pomace beverage (RG) or 150 ml/day of a control beverage (Placebo) for a 6-week period each. The two treatments will be separated by a 2-week wash-out period.

At the end of the run-in, wash-out, and both treatment periods, participants will undergo fasting blood samples to evaluate key metabolic parameters. After each treatment period (RG or placebo), a standardized meal (960 kcal, 18% protein, 30% fat, 52% carbohydrates) will be administered along with 150 ml of either the polyphenol-rich beverage or the control beverage, for postprandial metabolic evaluations.

At the end of both treatments, hepatic fat content, fasting and postprandial metabolic parameters, microbiota composition and continuos glucose monitoring will be assessed.

Energy intake and habitual dietary composition will be evaluated at the end of the run-in, and at 6 weeks after the start of each treatment period using a 7-day food diary.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >25 and ≤35 kg/m2
* Cholesterolemia ≤ 250 mg/dl and Triglyceridemia ≤ 200 mg/dl.
* type 2 Diabetes in good glycemic control (Hb1Ac ≤7.5%) treated with diet alone or diet + metformin.

Exclusion Criteria:

* Cardiovascular events (myocardial infarction and/or stroke)
* Renal insufficiency (serum creatinine >1.5 mg/dl) and liver failure (ALT/AST twice the normal values)
* Anemia (Hb <12 g/dl) or other chronic disease
* Insulin therapy and other hypoglycemic drugs other than metformin
* Habitual intense physical activity

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Differences in liver fat content | At baseline and at the end of 6 weeks of each treatment
  Differences in liver fat content after the intake of polyphenol rich drink (RGPD) for 6 weeks, as compared to Control drink (Placebo). Liver fat content will be assessed by magnetic resonance spectroscopy (MRI).

SECONDARY OUTCOMES:
Differences in glycemic variability | At baseline and at the end of 6 weeks of each treatment
  Differences in glycemic variability after the intake of polyphenol rich drink (RGPD) for 6 weeks, as compared to control drink (placebo). Glycemic variability will be assessed by Continuos Glucose Monitoring (CGM) during the 7 days before the end of each treatment.
Differences in glucose response | At the end of 6 weeks of each treatment
  Differences in fasting and postprandial plasma glucose response to a standard test meal at the end of the 6-week treatment with polyphenol rich drink (RGPD) as compared to control drink (placebo). Plasma glucose concentration will be assessed by enzymatic colorimetric methods.
Differences in insulin response | At the end of 6 weeks of each treatment
  Differences in fasting and postprandial plasma insulin response to a standard test meal at the end of the 6-week treatment with polyphenol rich drink (RGPD) as compared to control drink (placebo). Plasma insulin concentration will be assessed by ELISA method.
Differences in fasting lipid concentrations | At the end of 6 weeks of each treatment
  Differences in fasting plasma triglycerides, total cholesterol, HDL-cholesterol and LDL-cholesterol concentration at the end of the 6-week treatment with polyphenol rich drink (RGPD) as compared to control drink (placebo). Plasma lipid concentrations will be assessed by enzymatic colorimetric methods.
Differences in postprandial triglyceride response | At the end of 6 weeks of each treatment
  Differences in postprandial plasma triglycerides concentration at the end of the 6-week treatment with polyphenol rich drink (RGPD) as compared to control drink (placebo). Plasma triglyceride concentrations will be assessed by enzymatic colorimetric methods.
Differences in gastrointestinal hormones response | At the end of 6 weeks of each treatment
  Differences in fasting and postprandial plasma GLP-1, PYY and Ghrelin concentration at the end of the 6-week treatment with polyphenol rich drink (RGPD) as compared to control drink (placebo). Plasma concentrations of GLP-1, PYY and Ghrelin will be assessed by ELISA methods.
Differences in inflammatory markers | At the end of 6 weeks of each treatment
  Differences in fasting and postprandial serum hs-CRP concentration at the end of the 6-week treatment with polyphenol rich drink (RGPD) as compared to control drink (placebo). Serum concentrations of hs-CRP will be assessed by immunoturbidimetric method.
Differences in gut microbiota composition | At the end of 6 weeks of each treatment
  Differences in microbiota composition at the end of the 6-week treatment with polyphenol rich drink (RGPD) as compared to control drink (placebo). Microbiota analysis will be assessed on feacal samples by metagenomics.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalba Giacco, Senior Researcher, Principal Investigator — CNR; Luigi Russo, Senior Researcher, Study Director — CNR; Lutgarda Bozzetto, Full Professor, Principal Investigator — Federico II Univerisity
Locations (1):
- Federico II University, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol